CLINICAL TRIAL: NCT01893151
Title: A Randomized, Double-blind Study to Evaluate the Efficacy of Iguratimod Versus Placebo in Patients With Rheumatoid Arthritis on Magnetic Resonance Imaging (MRI)
Brief Title: Effectiveness of Iguratimod Versus Placebo to Treat Early Rheumatoid Arthritis on MRI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMM-3
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2013-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Iguratimod; MRI; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — iguratimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iguratimod (Experimental): Iguratimod:25 mg/tablet, taken orally, 2 tablets/day (bid),52week
  Interventions: Drug: Iguratimod
- Iguratimod placebo (Placebo Comparator): Iguratimod placebo:25 mg/tablet, taken orally, 2 tablets/day (bid),24week;Iguratimod:25 mg/tablet, taken orally, 2 tablets/day (bid),28week
  Interventions: Drug: Iguratimod placebo

INTERVENTIONS:
Drug: Iguratimod — Iguratimod placebo:25 mg/tablet, taken orally, 2 tablets/day (bid),52week
  Other Names: Iremod
  Arms: Iguratimod
Drug: Iguratimod placebo — Iguratimod placebo:25 mg/tablet, taken orally, 2 tablets/day (bid),24week; Iguratimod:25 mg/tablet, taken orally, 2 tablets/day (bid),28week.
  Arms: Iguratimod placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of Iguratimod versus placebo on synovial inflammation,bone erosion and bone edema as measured by MRI of wrist and Metacarpophalangeal joints in patients with early Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) is a powerful imaging modality that is now widely used in both scientific research and clinical settings to visualise joints of patients with RA. MRI is able to image structural damage and soft tissue changes, ie, synovitis, bone oedema, damage to cartilage and bone, as well as tendon pathology. MRI is more responsive to change in joint damage and can be used to monitor disease progression.

In this studly,MRI of the dominant wrist was performed at baseline ,24 weeks and at 52 weeks, using a 1.5T or 3.0T MRI with a dedicated high-resolution wrist phased array coil.The same scanner and wrist coil were used for three examinations. The hand was placed in the wrist coil at the patient's side with the coil anchored to the base tray to reduce motion artefacts. The MRI sequences in this study included the OMERACT recommended MRI core set of sequences.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of RA according to the diagnostic criteria of the American College of Rheumatology (ACR) (revised in 1987)
* Rheumatoid Arthritis for 3 months to 2 years from the time of the initial diagnosis
* Functional Class II-III
* Subjects have active RA at the time of screening
* Must have a negative Pregnancy test and use adequate method of contraception throughout the trial
* Must have at least 4 tender joints and 4 swollen joints(involved in DAS28) and among these,at least one swollen Metacarpophalangeal joint is essential
* Has a C-reactive protein ≥ 10 mg/L OR Erythrocyte Sedimentation Rate (ESR) ≥ 28 mm/hr
* Written informed consent

Exclusion Criteria:

* Preceding treatment with DMARDs, immunosuppressants (cyclophosphamide, cyclosporine, azathioprine, etc.), biological agents or tripterygium within 12 weeks prior to study entry
* Chest x-ray abnormalities, such as tuberculosis, interstitial pulmonary fibrosis, etc
* ALT >1.5×ULN, AST >1.5×ULN, Cr >135umol/L or Cr >1.5mg
* WBC<4×109/L，HGB<85g/L，PLT<100×109/L
* Subjects with serious cardiovascular, renal, hematologic,endocrine diseases or malignant
* Subjects with immunodeficiency, uncontrolled infection and active gastrointestinal disease
* Pregnant, intend to become pregnant, or are breastfeeding
* Subjects with other rheumatological diseases such as SLE, mixed connective tissue disease, scleroderma, polymyositis, etc
* Subjects with inflammatory arthritis, such as gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease
* Subjects with intra-articular corticosteroid injections within 6 weeks prior to study entry
* Allergic to any of the study drugs
* History of alcoholism
* Subjects with mental illness
* Subjects receiving live vaccines recently
* Subjects participating in other clinical study within 3 months prior to study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in RA magnetic resonance imaging scoring system (RAMRIS) | week 52
Change from baseline in modified Total Sharp Score (mTSS) | week 52
Percentage of patients with ACR 20 response | week 52
Change in Disease Activity as measured by the DAS28 | week 52

SECONDARY OUTCOMES:
Change from baseline in RAMRIS | week 24
Change from baseline in mTSS | week 24
Percentage of patients with ACR 20 response | week 10, week 24, week 40
Change from baseline in Disease Activity Score 28 (DAS28) | : week 10, week 24, week 40
Percentage of patients with ACR 50 response | week 10, week 24, week 40, week 52
Percentage of patients with ACR 70 response | week 10, week 24, week 40, week 52
Percentage of patients with Simplified Disease Activity Index (SDAI) ≤ 3.3 | week 10, week 24, week 40, week 52
Change from baseline in Simplified Disease Activity Index (SDAI) | week 10, week 24, week 40, week 52
Change from baseline in Health Assessment Questionnaire (HAQ) | week 10, week 24, week 40, week 52

CONTACTS AND LOCATIONS:
Overall Officials: Jieruo Gu, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital Of Sun Yat-sen University, Guangzhou, Guangdong, China